CLINICAL TRIAL: NCT06959394
Title: Comparison of the Effectiveness of Therapeutic Ultrasound and Phonophoresis Applications in Patients With Chronic Low Back Pain
Brief Title: Comparison of the Effectiveness of Therapeutic Ultrasound and Phonophoresis in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Mustafa Savaş Torlak, principle invastigator, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayMST
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — High-Energy Shock Waves; Phonophoresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US (Experimental): Participants will be treated with 1.5 W/cm2, 6 min (transmitting agent aquasonic gel) ultrasound.
  Interventions: Other: Ultrasound
- Phonophoresis (Experimental)
  Interventions: Other: Phonophoresis
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ultrasound — Participants will receive ultrasound at 1.5 W/cm2 for 6 minutes (transmitter agent aquasonic gel) 5 sessions per week for 2 weeks.
  Arms: US
Other: Phonophoresis — Participants will receive ultrasound with 1.5 W/cm2, 6 min (transmitter diclofenac gel) for 5 sessions per week for 2 weeks.
  Arms: Phonophoresis
Other: Placebo — Participants will receive 0 W/cm2, 6 min ultrasound, 5 sessions per week for 2 weeks.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects of therapeutic ultrasound and phonophoresis applications on pain, range of motion, flexibility and functional capacity in patients with chronic low back pain. The study is planned as the first scientific study comparing the effectiveness of these two physiotherapy methods in the treatment of chronic low back pain. It is aimed to make national and international publications with the data obtained at the end of the study.

The study will be conducted in a randomised single-blind, placebo-controlled design. 60 patients aged 18-30 years with chronic low back pain will be divided into 3 groups: therapeutic ultrasound (US) application, phonophoresis application and placebo US group. In addition to ultrasound and phonophoresis, TENS, infrared and low back exercises will be applied to all groups as treatment. Pain intensity (VAS), functional status (Oswestry disability index), flexibility (Sit-to-Sit test) and range of motion (goniometric measurements) will be assessed throughout the treatment period.

The study aims to make an important contribution from a clinical and economic point of view, given the increasing prevalence of low back pain worldwide and the need for treatment. The findings may guide the development of future treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

Individuals with low back pain for more than 3 months and pain intensity more than 5 according to VAS will be included in the study

Exclusion Criteria:

patients who have undergone surgical operations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pain severity | Baseline and after 2 weeks intervation
  Visual Analog Scale

SECONDARY OUTCOMES:
functional state | Baseline and after 2 weeks intervation
  Oswestry Disability Index
Flexibility | Baseline and after 2 weeks intervation
  Sit and Reach Test
range of motion of the joint | Baseline and after 2 weeks intervation
  Goniometry